CLINICAL TRIAL: NCT01019070
Title: Multiple-Dose Pharmacokinetics of BMS-650032 in Subjects With Hepatic Impairment Compared to Healthy Subjects
Brief Title: Hepatic Impaired Subjects Compared to Healthy Subjects Receiving Multi-dose BMS-650032
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI447-012
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMS-650032 in Child-Pugh A (Active Comparator)
  Interventions: Drug: BMS-650032
- BMS-650032 in Child-Pugh B (Active Comparator)
  Interventions: Drug: BMS-650032
- BMS-650032 in Child-Pugh C (Active Comparator)
  Interventions: Drug: BMS-650032
- BMS-650032 in Healthy Subjects (Active Comparator)
  Interventions: Drug: BMS-650032

INTERVENTIONS:
Drug: BMS-650032 — Capsules, Oral, 200 mg, BID, 7 Days

SUMMARY:
The purpose of this study is to assess the effects of hepatic impairment on the multiple dose pharmacokinetics of BMS-650032.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 70, with hepatic impairment conforming to Child-Pugh class A,B or C
* Each matched control subjects determined to be healthy

Exclusion Criteria:

* History of esophageal and gastric bleeding within the past 6 months
* Primarily cholestatic liver disease
* Active alcoholic hepatitis
* Stable encephalopathy of ≥Stage 2
* Presence of severe ascites or edema
* Presence of hepatopulmonary or hepatorenal syndrome
* Positive for HIV
* Positive for HCV, unless HCV RNA is undetectable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters including Cmax, Tmax,AUC(TAU),Vss/F, T-Half, CLT/F and AI | Day 10

SECONDARY OUTCOMES:
Assess the safety and tolerability of BMS-650032 in subjects with hepatic impairment and in healthy subjects. This will be measured by: blood chemistries, hematology, urinalysis and ECGs | Day 10
Assess the relationship between the Child-Pugh classification (including its components) and BMS-650032 PK parameters. This will be measured by frequent pharmacokinetics blood samples. | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Advanced Clinical Res Inst, Anaheim, California
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- [Derived] Eley T, He B, Chang I, Colston E, Child M, Bedford W, Kandoussi H, Pasquinelli C, Marbury TC, Bertz RJ. The effect of hepatic impairment on the pharmacokinetics of asunaprevir, an HCV NS3 protease inhibitor. Antivir Ther. 2015;20(1):29-37. doi: 10.3851/IMP2773. Epub 2014 Apr 7. PMID 24704773
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx